CLINICAL TRIAL: NCT00475137
Title: A Randomized, Single-Blind Comparison of Lamotrigine Add-on Versus Switch to Lamotrigine Monotherapy in the Treatment of Bipolar II Depression Unresponsive to Antidepressant Treatment
Brief Title: Lamotrigine Alone Compared to Lamotrigine Plus Antidepressant for the Treatment of Bipolar II Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H06-03732
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Bipolar II Disorder, Most Recent Episode Major Depressive
Keywords: Bipolar II Disorder; depression; Lamotrigine; Add On antidepressant; randomized; single blind; parallel group
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine Plus Antidepressant (Experimental): Subjects will be randomized to one of two study arms at baseline. Those in the first treatment arm will be prescribed lamotrigine in addition to the antidepressant medication they were prescribed prior to study entry.
  Interventions: Drug: Lamotrigine
- 2. Lamotrigine Monotherapy (Active Comparator): Subjects in the second treatment arm will discontinue their antidepressants and will be prescribed lamotrigine monotherapy. Lamotrigine will be initiated at 25mg daily for two weeks, then increased to 50mg daily for one week, and then increased to 100 mg daily. The dose may then be adjusted upward or downward by 50-100mg weekly, at the investigator's discretion, provided that it remains within the protocol defined range of 100mg - 400mg daily.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine will be initiated at 25mg daily for two weeks, then increased to 50mg daily for one week, and then increased to 100 mg daily. The dose may then be adjusted upward or downward by 50-100mg weekly, at the investigator's discretion, provided that it remains within the protocol defined range of 100mg - 400mg daily. For subjects in this combination therapy arm, antidepressant dose will remain constant throughout the study.
  Other Names: Lamictal
  Arms: Lamotrigine Plus Antidepressant
Drug: Lamotrigine — Lamotrigine will be initiated at 25mg daily for two weeks, then increased to 50mg daily for one week, and then increased to 100 mg daily. The dose may then be adjusted upward or downward by 50-100mg weekly, at the investigator's discretion, provided that it remains within the protocol defined range of 100mg - 400mg daily. Subjects in this group will discontinue their antidepressants prescribed to them before the study.
  Other Names: Lamictal
  Arms: 2. Lamotrigine Monotherapy

SUMMARY:
Depression is a medical condition characterized by feeling sad even when good things happen, having low energy and motivation, and sometimes even experiencing suicidal thoughts. Bipolar II Disorder is an illness in which periods of depression alternate with periods of abnormally elevated mood, energy and activity, referred to as hypomania. After Major Depressive Disorder, Bipolar II Disorder is the most common cause of depression. Unfortunately, antidepressant medications, used alone, do not work as well in treating Bipolar depression as they do in treating other kinds of depression. Lamotrigine is a medication which studies show is effective in treating Bipolar depression. The investigators will determine if lamotrigine works best to treat Bipolar II depression if it is used alone, or if it is taken with an antidepressant. In the first part of our investigation, people with Bipolar II depression who have not responded to an antidepressant will either add lamotrigine to their antidepressant, or will stop the antidepressant and take lamotrigine alone. They will see the study doctor for 6 visits over 8 weeks, and will answer questions about their depressive symptoms and their overall health. The purpose of this study phase is to determine which treatment works best to treat active Bipolar depression. In the second part of the study, people who have responded to their assigned treatment may continue to receive it for another 44 weeks. They will see the study doctor monthly, and will answer similar questions about their health. Participants will also receive a physical examination and get a blood test three times during the study. The purpose of the second phase is to ascertain which treatment is best at preventing relapses of depression. The investigators hypothesize that people who take Lamotrigine plus an antidepressant will recover from their depression more completely, have a longer period of wellness, and have better quality of life compared to those taking Lamotrigine alone.

DETAILED DESCRIPTION:
PURPOSE: To evaluate the efficacy and safety of lamotrigine when added to antidepressant medication, versus lamotrigine monotherapy, in the treatment and prevention of major depression in patients with Bipolar II Disorder which has not responded to antidepressant treatment alone.

HYPOTHESIS: Our primary hypothesis is that depressed patients with Bipolar II Disorder using lamotrigine plus antidepressant, as compared to those using lamotrigine monotherapy, will experience a greater decrease in their score on the Montgomery-Asberg Depression Rating Scale, a standard measure of severity of depression. The investigators also hypothesize that patients using lamotrigine in combination with antidepressant will have a greater survival time without experiencing depressed, manic, or hypomanic episodes during maintenance therapy, and an improved quality of life, compared to those receiving lamotrigine monotherapy.

JUSTIFICATION: Bipolar Disorder is a severe and recurrent psychiatric illness which is associated with high rates of mental health service utilization and functional disability. 15% - 20% of patients will complete suicide, the greatest rate of any psychiatric illness. With a lifetime prevalence of 3% - 5%, over one million Canadians suffer from this potentially disabling condition.

Bipolar I Disorder is characterized by one or more manic or mixed episodes, frequently in combination with episodes of depression. It has been well studied, and effective treatments are available for the depressed, manic, and maintenance phases of this condition. Bipolar II Disorder consists of periods of depression, plus one or more hypomanic (mild manic) episodes. The depressed phase of Bipolar II illness is overwhelmingly responsible for its substantial burden. Long-term follow-up studies demonstrate that patients experience depressive symptoms almost 40 times more often than symptoms of hypomania, and that even mild depressive symptoms are associated with significant functional impairment. Hypomanic episodes, conversely, are generally short, infrequent, and do not significantly impair functioning.

Bipolar II Disorder has been under-recognized, primarily due to its frequent misdiagnosis as Major Depressive Disorder. However, it is becoming increasingly clear that it is the most common Bipolar phenotype, affecting up to 80% of people with Bipolar illness. Underestimation of its prevalence has led to it being understudied. To date, no large randomized controlled trials exclusively involving Bipolar II patients have been published. Clinical decisions regarding the treatment of Bipolar II Disorder must therefore be extrapolated from research on Bipolar I patients, or based on the results of small open label studies. Clinical trials in Bipolar I samples show conclusively that mood stabilizing medications such as Lithium are the optimal treatment, and that antidepressant therapy may potentiate a switch into mania, or the development a rapid cycling course of illness. Several lines of evidence, however, including genetic, family, and long-term follow-up studies, suggest that Bipolar II Disorder is a distinct illness from Bipolar I Disorder. Making treatment decisions based on data from Bipolar I patients may therefore be inappropriate. While some open-label studies support the efficacy of mood stabilizing medications in Bipolar II Disorder, others suggest that Bipolar II patients may respond to antidepressant monotherapy. Antidepressants may be less effective in treating Bipolar II Disorder than Major Depressive Disorder, however, and Bipolar patients are over-represented in the treatment refractory population.

In clinical practice, combining an antidepressant and a mood stabilizing medication is a commonly used approach to treating Bipolar II depression. Lamotrigine is a mood stabilizing medication which has demonstrated efficacy in treating the depressed phase of Bipolar I Disorder, though not all studies have produced positive results. Therefore, the current study compares the efficacy and safety of the addition of lamotrigine to antidepressant medication, versus a switch of antidepressant to lamotrigine monotherapy, in the treatment of Bipolar II depression which has not responded to treatment with antidepressant medication.

OBJECTIVES: To evaluate the efficacy of lamotrigine in combination with antidepressant medication, versus lamotrigine monotherapy, over 8 weeks in the treatment of major depression in patients with Bipolar II Disorder. The investigators will also compare response and remission rates for depressive symptoms on a commonly-used metric of depression severity; effect on quality of life; level of patient acceptance; and safety and tolerability of the two treatment arms. A 44-week maintenance phase will assess the efficacy of the two treatment arms in preventing episodes of depression, mania, and hypomania.

RESEARCH METHOD: This is a randomized, single-blind, parallel-group study comparing the addition of lamotrigine to antidepressant medication, versus lamotrigine monotherapy, in the treatment of Bipolar II major depression. Approximately 100 patients will be randomized. During a screening phase, informed consent will be obtained, patient eligibility will be assessed, and previous psychoactive medications will be discontinued for a period of at least five half-lives. A baseline psychiatric assessment will be completed, including relevant clinical scales, physical examination, and protocol-required laboratory investigations. Patients who meet eligibility criteria will be enrolled in the study and randomized to one of the two treatment arms at the baseline visit. One study group will receive lamotrigine 100-400 mg daily plus antidepressant medication, while the other will receive lamotrigine 100-400 mg daily as monotherapy. Study visits will occur at baseline and at weeks 1, 2, 4, 6, and 8. Psychiatric status will be assessed by interview, and information regarding symptoms of depression and hypomania will be specifically obtained using clinical scales. Overall quality of life will be assessed at baseline and endpoint using a validated instrument. Adverse events, including mood switch into mania or hypomania, will be enumerated. Study endpoint will occur at week 8, or if the patient is withdrawn from the study due to non-response, adverse events, or for other reasons.

Subjects who meet the protocol-defined criteria for treatment response will be offered the opportunity to continue their assigned treatment during a 44-week maintenance study phase. Subjects will be assessed every 4 weeks during this study period. At each visit, information will be collected regarding symptoms of depression, mania or hypomania, overall psychiatric status, and adverse events. Medication adherence will be assessed at each visit. Assessment of quality of life, physical examination, and laboratory measures will be performed at endpoint.

SUMMARY: This is a 52 week study of the efficacy and safety of lamotrigine plus antidepressant, versus monotherapy with lamotrigine, in the treatment of major depression in patients with Bipolar II Disorder who have not responded to antidepressant treatment. The study has 4 phases: screening, enrollment, and acute treatment, and maintenance treatment.

Diagnosis of Bipolar II Disorder will be confirmed by clinical interview, according to DSM-IV-TR criteria. Presence and severity of depressive symptoms will be assessed with the Montgomery-Asberg Depression Rating Scale (MADRS). Subjects with confirmed Bipolar II Disorder,a MADRS score of at least 18, and no exclusion criteria, are eligible to participate in the study. Subjects who provide written informed consent will enter the screening phase. During the screening phase, demographic information including age, ethnicity, psychiatric and medical history, family psychiatric history, and previous medication trials will be collected. Vital signs and weight will be recorded, and blood work for hematology, serum chemistry, fasting glucose, thyroid function, urinalysis, urine toxicology, and pregnancy test, if appropriate, will be collected. A physical examination will be performed. Clinical rating scales will be administered, including the MADRS, the Young Mania Rating Scale (YMRS), and the Clinical Global Impression for Bipolar Disorder (CGI-BP) Severity and Change Scales. Psychotropic medications not allowed under the protocol will be tapered and discontinued for a period of at least 5 half-lives before the baseline visit. Subjects who continue to meet inclusion criteria after the screening phase will be randomized to study medication at the baseline visit. At the baseline visit, the above clinical rating scales will be readministered. Quality of life will be measured with the Quality of Life, Enjoyment, and Satisfaction Questionnaire (QLESQ).

Subjects will be randomized to one of two study arms at baseline. Those in the first treatment arm will be prescribed lamotrigine in addition to the antidepressant medication they were prescribed prior to study entry. Subjects in the second treatment arm will discontinue their antidepressants and will be prescribed lamotrigine monotherapy. Lamotrigine will be initiated at 25mg daily for two weeks,then increased to 50mg daily for one week, and then increased to 100 mg daily. The dose may then be adjusted upward or downward by 50-100mg weekly, at the investigator's discretion, provided that it remains within the protocol defined range of 100mg - 400mg daily. For subjects in the combination therapy arm, antidepressant dose will remain constant throughout the study. Treatment will be prescribed in an open-label fashion, but subjects will be assessed by an investigator who is blinded to treatment assignment.

Study visits for the acute treatment phase will occur at baseline, and at weeks 1, 2, 4, 6, and 8. At each visit, patients will undergo a review of study medications and other treatments, including pill counts. Adverse events will be recorded. Presence and severity of symptoms will be assessed at each visit via the MADRS, YMRS, and CGI-BP. Weight and vital signs will be measured at each visit. At study endpoint, quality of life will be reassessed with the QLESQ, and laboratory measures, including a serum pregnancy test, will be repeated. Endpoint will be reached at study week 8, or if the subject or the investigator withdraws the subject for any reason.

The primary outcome measure for the acute study phase will be change in severity of depressive symptoms, as determined by change in MADRS score from baseline to endpoint. Secondary outcomes will include rates of response to treatment (defined as 50% decrease in MADRS score); remission rates (defined as MADRS score <8); average time to response and remission; induction of mania or hypomania, as measured by change in YMRS scores (with hypomania defined as YMRS score >10 to 15 and mania defined as YMRS >16); rates of adverse events, as measured by patient report, and changes in vital signs, weight, and laboratory measures; improvement in quality of life, determined by change in QLESQ scores; and study completion rates.

Subjects who meet the criteria for remission at endpoint of the acute study phase will be offered the opportunity to continue their assigned treatment for a 44 week maintenance phase. The dosage of lamotrigine may be adjusted at the discretion of the investigator, but must remain in the range of 100-400 mg daily. No adjustments may be made in antidepressant dose in those subjects in the combination therapy arm. Study visits will occur every 4 weeks for 44 weeks. At each visit, MADRS, YMRS, and CGI-BP will be administered; weight and vital signs will be measured; adverse events will be recorded; and review of medications and pill counts will be performed. The QLESQ and laboratory measures will be repeated at endpoint. The primary outcome for the maintenance study phase will be survival time until the emergence of a depressed, manic, or hypomanic episode. Secondary outcome measures will include survival time in the study until withdrawal for any reason; frequency and severity of side effects; overall psychiatric status as determined by score on the CGI-BP; and quality of life, determined by QLESQ score.

Experimental aspects of the study include the use of lamotrigine and antidepressants for the treatment of depression in patients with Bipolar II Disorder, as neither medication is approved for this use by Canadian health authorities. While random assignment of patients to study groups may also be considered an experimental approach, both lamotrigine monotherapy and the combination of lamotrigine and antidepressant medication are commonly used approaches to treating Bipolar II Disorder in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible to participate in this trial:

1. Males or females, inpatients or outpatients, aged 17 to 70 years inclusive.
2. Diagnosis of Bipolar II Disorder, current episode depressed, without psychotic features. Specifically, patients must have experienced at least one previous episode of hypomania lasting at least 2 days, and no previous manic episodes.
3. The current episode of depression has a duration of at least 6 weeks.
4. Montgomery-Asberg Depression Rating Scale score of at least 18.
5. If female and of child-bearing age, must be using a reliable method of birth control. Reliable methods of birth control include: oral contraceptive pill or patch or surgically implanted device; intra-uterine device (IUD); tubal ligation; barrier device such as diaphragm or condom plus spermicidal jelly or foam; or abstinence.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible to participate in the trial:

1. Manic or hypomanic symptoms, defined as a YMRS score of 16 or greater.
2. Treatment with ECT or a depot antipsychotic medication within eight weeks prior to enrolment; or treatment with an experimental drug within 30 days prior to enrolment.
3. Known lack of response to, or intolerance for, Lamotrigine. Lack of response is defined as failure of depressive symptoms to improve after a trial of an acceptable dose of medication, ie. 100 mg daily or greater of Lamotrigine for at least four weeks.
4. Depressive symptoms secondary to substance use or a general medical condition, in the opinion of the investigator.
5. Diagnosis of an anxiety disorder, including Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Obsessive Compulsive Disorder, Specific Phobia, Post-Traumatic Stress Disorder, or Acute Stress Disorder, which was the primary focus of clinical attention in the year preceding enrolment.
6. Diagnosis of Schizophrenia, Schizoaffective Disorder, or Delusional Disorder.
7. Substance dependence within one month of enrolment, except for dependence in full remission, and except for caffeine or nicotine dependence, as defined by the DSM-IV-TR.
8. Diagnosis of Borderline Personality Disorder, Narcissistic Personality Disorder, Histrionic Personality Disorder, or Antisocial Personality Disorder, which was the primary focus of clinical attention in the year preceding enrolment.
9. Significant risk of harm to self or others, in the opinion of the investigator.
10. Use of any cytochrome P450 inducer or inhibitor within five half-lives prior to enrolment.
11. Pregnancy or lactation in female subjects.
12. Unstable or inadequately treated medical illness, as judged by the investigator.
13. Liver function tests (AST and ALT) three times the upper limit of normal.
14. Glomerular Filtration Rate (GFR) of less than 60 mL/min per 1.73m2
15. A history of significant cardiac conduction abnormalities, as determined by the investigator.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Lamotrigine monotherapy versus Lamotrigine plus antidepressant in the acute and maintenance treatment of Bipolar II depression as evidence by decrease in Montgomery-Asberg Depression Rating Scale (MADRS) score from baseline to endpoint. | 8 weeks

SECONDARY OUTCOMES:
Rates of response to treatment and remission in both treatment arms maintenance efficacy of treatments as evidenced by relapse rates. Rates of treatment associated mania or hypomania as evidenced by increased score on the Young Mania Rating Scale (YMRS). | 44 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Bond, MD, Principal Investigator — University of British Columbia; Lakshmi Yatham, MD, Study Director — University of British Columbia; Edwin Tam, MD, Study Director — University of British Columbia; Mauricio Kunz, Dr., Study Director — University of British Columbia; Kyooseob Ha, Dr., Study Director — Seoul National University Bundang Hospital; Wetid Pratoomsri, Dr., Study Director — Chachoengsao Hospital Thailand
Locations (1):
- University of British Columbia Mood Disorders Centre, Vancouver, British Columbia, Canada